CLINICAL TRIAL: NCT05211895
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Multicentre, International Study of Durvalumab Plus Domvanalimab(AB154) in Participants With Locally Advanced (Stage III), Unresectable Non-small Cell Lung Cancer Whose Disease Has Not Progressed Following Definitive Platinum-based Concurrent Chemoradiation Therapy
Brief Title: A Global Study to Assess the Effects of Durvalumab + Domvanalimab Following Concurrent Chemoradiation in Participants With Stage III Unresectable NSCLC
Acronym: PACIFIC-8
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9075C00001; 2021-004327-32 (EudraCT Number)
Record Dates: First submitted 2022-01-11; First posted 2022-01-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; locally advanced; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Durvalumab + Domvanalimab (Experimental): Durvalumab and domvanalimab as an IV infusion q4w, starting on Day 1 for up to a maximum of 12 months
  Interventions: Drug: Durvalumab; Drug: Domvanalimab
- Arm B: Durvalumab + Placebo (Active Comparator): Durvalumab + placebo as an IV infusion q4w starting on Day 1 for up to a maximum of 12 months
  Interventions: Drug: Durvalumab; Other: Placebo

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (Intravenous infusion)
Drug: Domvanalimab — Domvanalimab IV (Intravenous infusion)
  Arms: Arm A: Durvalumab + Domvanalimab
Other: Placebo — Placebo IV (Intravenous infusion)
  Arms: Arm B: Durvalumab + Placebo

SUMMARY:
This is a Phase III, randomised, double-blind, placebo-controlled, multicentre, international study assessing the efficacy and safety of durvalumab (MEDI4736) and domvanalimab (AB154) compared with durvalumab plus placebo in adults with locally advanced (Stage III), unresectable NSCLC whose disease has not progressed following definitive platinum-based cCRT.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Participant must be ≥ 18 years at the time of screening.
2. Histologically- or cytologically-documented NSCLC and have been treated with concurrent CRT for locally advanced, unresectable (Stage III) disease
3. Provision of a tumour tissue sample obtained prior to CRT
4. Documented tumour PD-L1 status ≥ 1% by central lab
5. Documented EGFR and ALK wild-type status (local or central).
6. Patients must not have progressed following definitive, platinum-based, concurrent chemoradiotherapy
7. Participants must have received at least 2 cycles of platinum-based chemotherapy concurrent with radiation therapy
8. Participants must have received a total dose of radiation of 60 Gy ±10% (54 Gy to 66 Gy) as part of the chemoradiation therapy, to be randomised. Radiation therapy should be administered by intensity modulated RT (preferred) or 3D-conforming technique.
9. WHO performance status of 0 or 1 at randomization
10. Adequate organ and marrow function

EXCLUSION CRITERIA:

1. History of another primary malignancy, except for:

   * Malignancies treated with curative intent and adequate follow-up with no known active disease and have not required active treatment within the past 3 years before the first dose of study intervention and of low potential risk of recurrence.
   * Adequately resected non melanoma skin cancer or lentigo maligna without evidence of disease .
   * Adequately treated carcinoma in situ, including Ta tumors without evidence of disease.
2. Mixed small cell and non-small cell lung cancer histology.
3. Participants who receive sequential (not inclusive of induction) chemoradiation therapy for locally advanced (Stage III) unresectable NSCLC.
4. Participants with locally advanced (Stage III) unresectable NSCLC who have progressed during platinum-based cCRT.
5. Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy (excluding alopecia).
6. Participants with ≥ grade 2 pneumonitis from prior chemoradiation therapy.
7. History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, or idiopathic pneumonitis - regardless of time of onset prior to randomisation. Evidence of active non-CRT induced pneumonitis (≥ Grade 2), active pneumonia, active ILD, active or recently treated pleural effusion, or current pulmonary fibrosis
8. Active or prior documented autoimmune or inflammatory disorders (with exceptions)
9. Active EBV infection, or known or suspected chronic active EBV infection at screening
10. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2028-07-12 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 8 years after randomization
  Defined as time from randomisation until progression per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR), or death due to any cause in participants with PD-L1 TC ≥ 50%.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 8 years after randomization
  Defined as time from randomisation until progression per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR), or death due to any cause in participants with PD-L1 TC ≥ 1%
Overall Survival (OS) | Approximately 8 years after randomization
  Overall Survival (OS)
Objective Response Rate (ORR) | Approximately 8 years after randomization
  Objective Response Rate (ORR) per RECIST 1.1 as assessed by BICR
Duration of Response (DoR) | Approximately 8 years after randomization
  Duration of Response (DoR) using BICR assessment according to RECIST 1.1
Time from randomization to second progression (PFS2) | Approximately 8 years after randomization
  Time from randomization to second progression (PFS2)
Time from randomization to first date of distant metastasis or death (TTDM) | Approximately 8 years after randomization
  Time from randomization until the first date of distant metastasis or death in the absence of distant metastasis (TTDM).
Time to first subsequent therapy (TFST) | Approximately 8 years after randomization
  Time to first subsequent therapy (TFST)
Concentration of Durvalumab and Domvanalimab | Approximately 12 weeks after last IP dose
  The pharmacokinetics (PK) of Durvalumab and Domvanalimab as determined by concentration
PFS6, PFS12, PFS18, PFS24 | Approximately 6, 12, 18 and 24 months after randomization
  PFS at 6, 12, 18 and 24 months (proportion per Kaplan-Meier)
Anti-Drug Antibodies (ADAs) | Approximately 12 weeks after last IP dose.
  The immunogenicity of Durvalumab and domvanalimab as assessed by presence of Anti-Drug Antibodies (ADAs)
Time to deterioration in pulmonary symptoms (TTFCD) | Approximately 8 years after randomization
  Time to deterioration in pulmonary symptoms (TTFCD)
PFS investigator | Up to 8 years after randomization
  Defined as time from randomisation until progression per RECIST 1.1 as assessed by Investigator or death due to any cause in participants
OS 24 | Approximately 24 months after randomization
  Overall Survival (OS) at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Hidehito Horinouchi, MD, PhD, Principal Investigator — National Cancer Center Hospital; Alexander Spira, MD, PhD, Principal Investigator — Virginia Cancer Specialists Research Institute; Jinming Yu, MD, PhD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (224):
- United States (40):
  - Research Site, Chandler, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Fountain Valley, California
  - Research Site, Santa Rosa, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, Macon, Georgia
  - Research Site, Elmhurst, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Naperville, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Reno, Nevada
  - Research Site, East Brunswick, New Jersey
  - Research Site, Florham Park, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Johnson City, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Fort Sam Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Arlington, Virginia
  - Research Site, Fort Belvoir, Virginia
  - Research Site, Spokane Valley, Washington
  - Research Site, Appleton, Wisconsin
- Belgium (6):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Haine-Saint-Paul
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Sint-Niklaas
- Brazil (8):
  - Research Site, Barretos
  - Research Site, Londrina
  - Research Site, Porto Alegre
  - Research Site, Porto Velho
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Taubaté
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
- Chile (4):
  - Research Site, Las Condes
  - Research Site, Port Montt
  - Research Site, Santiago
  - Research Site, Temuco
- France (12):
  - Research Site, Aix-en-Provence
  - Research Site, Angers
  - Research Site, Bobigny
  - Research Site, Clermont-Ferrand
  - Research Site, Lille
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Quimper
  - Research Site, Saint-Grégoire
  - Research Site, Saint-Quentin
  - Research Site, Vantoux
  - Research Site, Villeurbanne
- Germany (19):
  - Research Site, Berlin
  - Research Site, Berlin-Zehlendorf
  - Research Site, Braunschweig
  - Research Site, Chemnitz
  - Research Site, Cologne
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Georgsmarienhütte
  - Research Site, Giessen
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Homburg
  - Research Site, Koblenz
  - Research Site, Krefeld
  - Research Site, Löwenstein
  - Research Site, Moers
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Tübingen
- Greece (3):
  - Research Site, Athens
  - Research Site, Holargos, Athens
  - Research Site, Thessaloniki
- Research Site, Hong Kong, Hong Kong
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Deszk
  - Research Site, Győr
  - Research Site, Salgótarján
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
- India (13):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Gūrgaon
  - Research Site, Howrah
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Marg Jaipur
  - Research Site, Mohali
  - Research Site, Namakkal
  - Research Site, New Delhi
  - Research Site, Varanasi
- Italy (4):
  - Research Site, Bergamo
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Udine
- Japan (17):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hidaka-shi
  - Research Site, Hirosaki-shi
  - Research Site, Itabashi-ku
  - Research Site, Kashihara-shi
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Sunto-gun
  - Research Site, Tokyo
  - Research Site, Yokohama
- Malaysia (4):
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
- Mexico (9):
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Monterrey
  - Research Site, Oaxaca City
  - Research Site, San Pedro Garza García
  - Research Site, Sonora
  - Research Site, Veracruz
- Norway (4):
  - Research Site, Bodø
  - Research Site, Gjøvik
  - Research Site, Oslo
  - Research Site, Trondheim
- Philippines (6):
  - Research Site, Bacolod
  - Research Site, City of Muntinlupa
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gliwice
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zielona Góra
- Romania (8):
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Floreşti
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Sibiu
  - Research Site, Suceava
  - Research Site, Timișoara
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, eManzimtoti
  - Research Site, Johannesburg
  - Research Site, Parktown
  - Research Site, Pretoria
- South Korea (6):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Jinju
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (6):
  - Research Site, Bilbao (Vizcaya)
  - Research Site, Castellon
  - Research Site, Córdoba
  - Research Site, El Palmar
  - Research Site, Palma de Mallorca
  - Research Site, Sabadell (Barcelona)
- Switzerland (3):
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Lausanne
- Taiwan (6):
  - Research Site, Hsinchu
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Hat Yai
- Turkey (Türkiye) (8):
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Çankaya
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Konya
- United Kingdom (11):
  - Research Site, Birmingham
  - Research Site, Brighton
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Cheltenham
  - Research Site, Edinburgh
  - Research Site, High Heaton/Newcastle Upon Tyn
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Truro
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- See also: 1-844-432-3892 Lung Cancer Study Locator details to CT.gov for the US sites only — https://www.lungcancerstudylocator.com/trial/listing/331601